CLINICAL TRIAL: NCT03714321
Title: Mechanical Insufflation-Exsufflation Compared With CPAP in Patients Admitted to an Intermediate Care Unit With Pneumonia: a Randomised Controlled Study.
Brief Title: Mechanical Insufflation-Exsufflation Compared With CPAP in Patients Admitted to an Intermediate Care Unit With Pneumonia
Acronym: CoughAssist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Fredrikke Christie Knudtzen, Specialist Registrar, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-20130102/j.nr. 2008-58-0035
Record Dates: First submitted 2018-10-10; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Pneumonia
Keywords: mechanical insufflation-exsufflation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Randomized non-blinded controlled pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical insufflation-exsufflation arm (Experimental): MIE will be given as prescribed by physician responsible at the intermediate care unit, typically every 4 hours. MIE will be administered with standard settings of insufflation 20 cm H2O and exsufflation 20 cm H2O, with possible individual changes from 10/-10 H2O up to 40/-40 H2O, and oxygen flow up to 15 l/min. The standard settings will be set to five cycles of 2 seconds insufflation, 3 seconds exsufflation with a three second pause between each cycle. Every treatment session consists of five rounds of five cycles, in all 25 insufflation/exsufflation, with time between each cycle of 30 seconds, meant used for suction.
  Interventions: Device: Mechanical insufflation-exsufflation (MIE)
- CPAP arm (No Intervention): CPAP will be given as prescribed by the physician responsible at the intermediate care unit, typically every 4 hours. CPAP will be administered with standard settings of H2O and an oxygen flow of 15L/min.

INTERVENTIONS:
Device: Mechanical insufflation-exsufflation (MIE) — Randomization of 30 patients, 15 in each arm, to receive either CPAP or MIE.
  Other Names: NIPPY Clearway
  Arms: Mechanical insufflation-exsufflation arm

SUMMARY:
Pneumonia, an infection in the lower airways, is a common cause of hospital contacts and a leading cause of death from infections worldwide. Pneumonia is treated with antibiotics, and while waiting for the effect thereof patients may need supportive treatment to help their lungs work optimally.

When patients suffering from pneumonia have problems breathing, Continuous Positive Airway Pressure (CPAP) is widely used. CPAP works by forcing air down the patient's airway. In patients with pneumonia, though CPAP has proven to provide more oxygen to the lungs compared to a standard oxygen mask, it does not have any effect on the outcome.

Mechanical insufflation-exsufflation (MIE), examined in this study, is given through a machine connected to a mask. If provides a positive airway pressure like CPAP, but the inwards pressure is followed immediately by a negative pressure forcing air and mucus up from the lower airways. MIE is currently used successfully in patients suffering from neuromuscular diseases. In these patients, MIE has shown to prevent hospital admission, prolong survival and delay time until need of permanent ventilation. There exists no studies examining the effect of MIE on patients with pneumonia without neuromuscular disorders.

The investigators therefore wish to study patients with severe pneumonia, admitted to an intermediate care unit, and compare patients treated with MIE to patients treated with CPAP.

30 patients will be included and randomly selected to receive either CPAP or MIE. They will be monitored through registration of oxygen need (liters/min) and oxygen levels, respiratory rate and the daily number of suction due to mucus.

Data from each patient regarding their age, sex, other known diseases, the severity of pneumonia, chest X-ray findings, antibiotic treatment up to and during the admission, days admitted, hours admitted to the intermediate care unit, if they are transferred to the intensive care unit and put on a ventilator, 30-days mortality and re-admittance within 30 days of being discharged, will be registered. To enter the study, the patients have to be 18 years old, able to sign a written consent form, have no current chest tube, no recent collapsed lung and no chronic lung disease.

The hypothesizes is that patients receiving MIE will be helped with coughing up mucus in the lower airways, and therefore have less need of oxygen, and that the patients receiving MIE will have a reduced risk of being transferred to the intensive care unit to receive ventilator support and spend shorter time in the intermediate care unit compared with the other group.

DETAILED DESCRIPTION:
Background

Mechanical insufflation-exsufflation (MIE) was invented to help mobilize secretion from the lower respiratory tract by simulating a cough [1]. It is widely used in patients who have neuromuscular disease and therefore reduced cough strength, both during hospital admissions, and in patients' homes. Delivered by a Cough Assistor device through a mask, MIE functions by delivering a positive inspiratory pressure followed immediately by a negative expiratory pressure [1].

In patients with neuromuscular disease, MIE prevents hospital admissions, improves survival rates and delay time to tracheostomy [1]. In this patient group, MIE has proven to be safe with few adverse effects, and generally well tolerated [1-3].

In patients with neuromuscular disease and an acute respiratory-tract infection, MIE in combination with non-invasive ventilation (NIV) is superior to NIV alone in removing secretion from the airways in patients with respiratory tract infections [2]. In a study among patients with severe chronic obstructive pulmonary disease (COPD) and difficulties clearing airway secretions after acute respiratory failure, MIE had a significant effect on both oxygenation and dyspnea [3].

Pneumonia is, with a yearly incidence of 5-11 per 1.000 adult population, a leading cause of morbidity worldwide [4]. Around 22-42% of adults with community-acquired pneumonia (CAP) require hospitalization [4]. Globally, pneumonia is the leading cause of death due to infections, and the mortality among hospitalized patients with pneumonia is 5.7-14% [4,5]. Pneumonia is seen with increased incidence in high risk patient groups such as the elderly, smokers, patients with immunodeficiencies and co-morbidities [6]. Early initiation of appropriate antimicrobial therapy is the cornerstone in treatment of pneumonia and has been shown to shorten the course of disease and lessen the risk of complications and mortality [7].

In the acute phase of the disease, in addition to effective antimicrobial treatment, supportive treatment is important to optimize the respiratory care of the patients. Continuous positive airway pressure (CPAP) delivered through a face mask is widely used as supportive treatment and improves oxygenation in patients with acute hypoxemic respiratory failure compared to oxygen delivered by mask [8]. CPAP also improves oxygenation in patients with pneumonia in a hospital setting compared to oxygen therapy, but the effect quickly resolves after discontinuation, and CPAP has failed to show effect on endotracheal intubation rate, hospital mortality and length of intensive care unit stay in patients with acute respiratory failure [8-10].

There are, to the investigators knowledge, no published studies who evaluate the effect of MIE on patients with acute respiratory-tract infections without neuromuscular disease.

The aim of this study is to investigate the safety and effect of MIE on patients hospitalized due to lower respiratory-tract infections and examine their outcome with the current standard treatment of CPAP.

Hypothesis Patients receiving MIE have better mobilization of secretions from the lower airways, and thereby faster oxygenation. Patients in the MIE group will have less need of ventilator support, and have a shorter admission to the intermediate care unit.

Methods

Study design This randomized clinical pilot study is conducted at the intermediate care unit at the Department of Infectious Diseases, Odense University Hospital, Denmark. The intermediate care unit consists of 3 beds, all served by a nurse with special training in intermediate care. Continuous monitoring of blood pressure, pulse, oxygen saturation and respiratory rate is available. The assessment of the patient and admittance to the intermediate care unit is determined by the senior infectious disease doctor on call.

Randomization In total, 30 patients will be included and undergo 1:1 randomization to receive either CPAP or CPAP followed by MIE.

Interventions CPAP will be administered through MR 810 (Fisher & Paykel Healthcare, Auckland, New Zealand) with standard settings of H2O and an oxygen flow of 15L/min [11]. CPAP is given by trained physiotherapists or nurses at the intermediate care unit.

MIE will be administered through the NIPPY Clearway (B&D Electromedical, Stratford-Upon-Avon, Warwickshire, United Kingdom) with standard settings of insufflation 20 cm H2O and exsufflation 20 cm H2O, with possible individual changes from 10/-10 H2O up to 40/-40 H2O, and oxygen flow up to 15 l/min [12]. The standard settings will be set to five cycles of 2 seconds insufflation, 3 seconds exsufflation with a three second pause between each cycle. Every treatment session consists of five rounds of five cycles, in all 25 insufflation/exsufflation, with time between each cycle of 30 seconds, meant used for suction. The MIE is given by trained physiotherapists or nurses at the intermediate care unit.

Clinical data The following data will be registered for each patient: age, sex, comorbidities, the severity of pneumonia using the CURB-65 score [13], chest radiograph findings, antibiotic treatment up to and during the admission, days of admission, hours admitted to the semi-intensive unit, transfer to intensive care unit (ICU), intubation and mechanical ventilation, in-hospital and 30-days mortality and re-admittance within 30 days of discharge. During the admission in the intermediate care unit, number of CPAP and MIE treatments, oxygenation and oxygen need (liters/min) every 2 hours for the first 24 hours, hereafter every 4 hours, respiratory rate every 6 hours for the first 24 hours, hereafter every day, and the daily number of suction in pharynx or trachea in each patient will be registered.

Paraclinical data For each patient, microbial growth from blood and sputum cultures will be registered, as will Polymerase Chain Reaction (PCR) results from sputum samples and relevant bacterial serology during admission, C-reactive protein (CRP), white blood cell count (WBC) and urea at time of admission, time of entering the intermediate care unit, time of discharge from the intermediate care unit and time of discharge from the hospital.

Statistical analysis Fisher's exact test and Wilcoxon rank sum will be used for categorical and continuous variables, respectively. A p-value of < 0.05 is considered statistically significant. The statistical analyses will be performed using STATA version 13.0.

ELIGIBILITY:
Inclusion Criteria:

* Community acquired or nosocomial pneumonia, diagnosed by new infiltrate on an x-ray chest and symptoms and/or objective findings acute lower airway infection
* 18 years or older
* able to participate in CPAP treatment 10 cm H2O for 5 minutes
* able to provide written consent

Exclusion Criteria:

* pneumothorax less than 4 weeks prior to admission
* current pleural tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-10-09 (Actual); Study Completion 2015-10-09 (Actual)

PRIMARY OUTCOMES:
Admission time in intermediate care unit | Admission to intermediate care unit (expected approx. 3-5 days)
  Time (in hours) of each patient spent admitted to the intermediate care unit
Need of mechanical ventilation | From admission to discharge/death, in the department responsible for the study, the mean duration of admittance is 7 days. Need of ventilation will be registered by investigator through review of patient chart after discharge from hospital.
  For each patient; any need of mechanical ventilation (yes/no) during the entire hospital admission in which the patient is included in the study.

SECONDARY OUTCOMES:
Oxygenation therapy | During the entire admission to the intermediate care unit (expected to be approx. 3-5 days) oxygen therapy will be registered every 2 hours for the first 24 hours of admittance, and every 4 hours thereafter until discharge.
  Registration of oxygen therapy (L/min)
Oxygenation saturation | During the entire admission to the intermediate care unit (expected to be approx. 3-5 days) oxygen saturation will be registered every 2 hours for the first 24 hours of admittance, and every 4 hours thereafter until discharge.
  Registration of oxygen saturation (%)
Respiratory rate | Registered at admission to the intermediate care unit, every 6th hour for the first 24 hours thereafter, and every 24 hours for the duration of admission to the intermediate care unit (approx.3-5 days).
  Registration of respiratory rate (number/minute) every 6th hours
Need of suction | During the entire admission to the intermediate care unit (approx.3-5 days), every episode of suction will be registered by the treating nurse, and total number of episodes will be registered every 24th hours until discharge.
  Registration of every episode of suction (number/day) and from which part of the airway (mouth, pharynx, trachea)
Treatment related adverse events | Registered daily on patient chart forms during entire admission to the intermediate care unit, and orally reported to the principal investigator during the admissions (approx. 3-5 days per patient).
  Registration of discontinuation of MIE, change in settings in MIE due to discomfort, reported adverse events after treatment. Registered in patient charts and/or reported by treating nurses/physiotherapists to principal investigator during patient admissions. No structural form used.

CONTACTS AND LOCATIONS:
Overall Officials: Isik Johansen, Prof., Principal Investigator — Odense University Hospital

IPD SHARING:
Plan to Share IPD: Undecided
No current plan for IPD sharing, will be reconsidered when we have decided if the pilot project will be expanded.

REFERENCES:
- [Background] Ellison RT III, Donowitz GR. Acute pneumonia. In: Bennett JE, Dolin R, Blaser MJ. Mandell, Douglas, and Bennett's Principles and Practice of Infectious Diseases. 8th Edn. Philadelphia, Elsevier Saunders, 2015; pp. 829-831.
- [Result] Homnick DN. Mechanical insufflation-exsufflation for airway mucus clearance. Respir Care. 2007 Oct;52(10):1296-305; discussion 1306-7. PMID 17894900
- [Result] Chatwin M, Simonds AK. The addition of mechanical insufflation/exsufflation shortens airway-clearance sessions in neuromuscular patients with chest infection. Respir Care. 2009 Nov;54(11):1473-9. PMID 19863831
- [Result] Winck JC, Goncalves MR, Lourenco C, Viana P, Almeida J, Bach JR. Effects of mechanical insufflation-exsufflation on respiratory parameters for patients with chronic airway secretion encumbrance. Chest. 2004 Sep;126(3):774-80. doi: 10.1378/chest.126.3.774. PMID 15364756
- [Result] Lim WS, Baudouin SV, George RC, Hill AT, Jamieson C, Le Jeune I, Macfarlane JT, Read RC, Roberts HJ, Levy ML, Wani M, Woodhead MA; Pneumonia Guidelines Committee of the BTS Standards of Care Committee. BTS guidelines for the management of community acquired pneumonia in adults: update 2009. Thorax. 2009 Oct;64 Suppl 3:iii1-55. doi: 10.1136/thx.2009.121434. No abstract available. PMID 19783532
- [Result] Welte T. Risk factors and severity scores in hospitalized patients with community-acquired pneumonia: prediction of severity and mortality. Eur J Clin Microbiol Infect Dis. 2012 Jan;31(1):33-47. doi: 10.1007/s10096-011-1272-4. Epub 2011 May 1. PMID 21533875
- [Result] Blasi F, Garau J, Medina J, Avila M, McBride K, Ostermann H; REACH study group. Current management of patients hospitalized with community-acquired pneumonia across Europe: outcomes from REACH. Respir Res. 2013 Apr 15;14(1):44. doi: 10.1186/1465-9921-14-44. PMID 23586347
- [Result] Delclaux C, L'Her E, Alberti C, Mancebo J, Abroug F, Conti G, Guerin C, Schortgen F, Lefort Y, Antonelli M, Lepage E, Lemaire F, Brochard L. Treatment of acute hypoxemic nonhypercapnic respiratory insufficiency with continuous positive airway pressure delivered by a face mask: A randomized controlled trial. JAMA. 2000 Nov 8;284(18):2352-60. doi: 10.1001/jama.284.18.2352. PMID 11066186
- [Result] Cosentini R, Brambilla AM, Aliberti S, Bignamini A, Nava S, Maffei A, Martinotti R, Tarsia P, Monzani V, Pelosi P. Helmet continuous positive airway pressure vs oxygen therapy to improve oxygenation in community-acquired pneumonia: a randomized, controlled trial. Chest. 2010 Jul;138(1):114-20. doi: 10.1378/chest.09-2290. Epub 2010 Feb 12. PMID 20154071
- [Result] Brambilla AM, Aliberti S, Prina E, Nicoli F, Del Forno M, Nava S, Ferrari G, Corradi F, Pelosi P, Bignamini A, Tarsia P, Cosentini R. Helmet CPAP vs. oxygen therapy in severe hypoxemic respiratory failure due to pneumonia. Intensive Care Med. 2014 Jul;40(7):942-9. doi: 10.1007/s00134-014-3325-5. Epub 2014 May 10. PMID 24817030
- [Result] MR810 technical manual. file:///C:/Users/lege4/Downloads/9e551a10-ef64-4514-a1bf-ce17cf08451e.pdf Date last accessed: July 12th 2017.
- [Result] NIPPY Clearway user manual. http://nippyventilator.com/wp-content/uploads/2016/02/2007v5-February2015-Clearway-IFU-English.pdf Date last updated: February 2015. Date last accessed: July 12th 2017.
- [Result] Lim WS, van der Eerden MM, Laing R, Boersma WG, Karalus N, Town GI, Lewis SA, Macfarlane JT. Defining community acquired pneumonia severity on presentation to hospital: an international derivation and validation study. Thorax. 2003 May;58(5):377-82. doi: 10.1136/thorax.58.5.377. PMID 12728155